CLINICAL TRIAL: NCT02664766
Title: Effects of Long-term Exercise on Psychological, Physiological, Biochemical and Alcohol-related Parameters in Heavy Drinkers
Brief Title: Effects of Long-term Exercise on Various Parameters in Heavy Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: European Social Fund (Other)
Responsible Party: Principal Investigator, Athanasios Z. Jamurtas, Dr, University of Thessaly
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UThessaly 2
Record Dates: First submitted 2016-01-18; First posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Heavy Drinking; Alcohol Abuse; Alcohol Use Disorder
Keywords: Heavy drinking; Heavy drinking cessation; Alcohol abuse; alcohol use disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control condition (No Intervention): Control condition with no intervention. Participants will be recording their daily alcohol consumption. No lifestyle modification during this period.
- Exercise training program (Experimental): Supervised 8-week exercise training program. Aerobic exercise (walking, jogging) of increasing duration at 50-60% HRR, at least two sessions per week.
  Interventions: Behavioral: Exercise training program

INTERVENTIONS:
Behavioral: Exercise training program — Supervised 8-week exercise training program. Aerobic exercise (walking, jogging) of increasing duration at 50-60% HRR, at least two sessions per week. Participants will be recording their daily alcohol consumption. Participants will also undergo three trials of acute exercise (before, at the 4th week and at the 8th week of exercise training) in order to investigate whether exercise training can lead to changes in acute responses to exercise. Each trial involves 30 min of exercise on a cycle ergometer at 50-60% HRR.
  Arms: Exercise training program

SUMMARY:
The purpose of this research is to examine the effects of long-term aerobic exercise of moderate intensity on psychological, physiological, biochemical, physiological and alcohol-related parameters in heavy drinkers, in order to investigate possible biochemical mechanisms by which exercise may be a healthy alternative to alcohol abuse.

DETAILED DESCRIPTION:
The mechanism of incentives that lead people to unhealthy habits such as excessive alcohol consumption is not only social, personal, and psychological, but also associated with neurochemical and neurobiological mechanisms.

Several programs have been developed to stop excessive drinking, but the success rates are small, while the relapse rates are very high, reaching up to 90%. Although there is some evidence for the beneficial effects of exercise on alcohol use disorders, research is limited. The present study investigates whether exercise can act as adjunct therapy for alcohol abuse cessation.

One of the basic assumptions is that the appropriate form of exercise in alcoholics will contribute to the secretion of beta-endorphin, which in combination with psychological pleasure, vitality, change of mood, reduced stress, increased confidence, and the shift of attention will help people to follow healthy lifestyles and abhor alcohol.

The research project is divided in three phases. In the first phase, the effect of acute exercise in critical psychological, physiological, biochemical and alcohol-related parameters associated with excessive alcohol consumption will be examined. In the second phase (current study), a long-term exercise program in conjunction with psychological support strategies aimed at alcohol abuse cessation will be developed, implemented and evaluated. Finally, in the third phase, based on the results of the previous phases, awareness programs in adolescent and adult populations will be designed and implemented as well as the dissemination of results and evaluation of the project will take place.

ELIGIBILITY:
Inclusion Criteria:

* Men drinking >14 drinks/week or >4 drinks/occasion; Women drinking >7 drinks/week or >4 drinks/occasion (1 drink = 14 grams of pure alcohol; definition of the NIAAA for drinking at low risk for developing an AUD; NIAAA, 2014)
* Individuals drinking 5 or more drinks on the same occasion on each of 5 or more days in the past 30 days (1 drink = 14 grams of pure alcohol; definition of the Substance Abuse and Mental Health Services Administration for heavy drinking; NIAAA, 2014) Alcohol Use Disorders Identification Test (AUDIT) score>8

Exclusion Criteria:

* Medical conditions or medication use that would preclude participation in aerobic exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes in alcohol consumption (grams of alcohol consumed weekly) | At baseline and at 4th week of control condition; at baseline (before intervention), at 4th week and at 8th week of intervention
  Self-recorded
Changes in Beta-endorphin levels | At baseline and at 4th week of control condition; at baseline (before intervention), at 4th week and at 8th week of intervention
  Measured by radioimmunoassay (RIA)

SECONDARY OUTCOMES:
Urge to drink | At baseline and at 4th week of control condition; at baseline (before intervention), at 4th week and at 8th week of intervention
  According to questionnaire
Cortisol | At baseline and at 4th week of control condition; at baseline (before intervention), at 4th week and at 8th week of intervention
  Measured by radioimmunoassay (RIA)
Adrenocorticotrophic hormone (ACTH) | At baseline and at 4th week of control condition; at baseline (before intervention), at 4th week and at 8th week of intervention
  Measured by radioimmunoassay (RIA)
Catecholamines (epinephrine, norepinephrine, dopamine) | At baseline and at 4th week of control condition; at baseline (before intervention), at 4th week and at 8th week of intervention
  Measured by radioimmunoassay (RIA)
C-reactive protein (CRP) | At baseline and at 4th week of control condition; at baseline (before intervention), at 4th week and at 8th week of intervention
  Semi-quantitative estimation with CRP Latex test kit
Complete blood count | At baseline and at 4th week of control condition; at baseline (before intervention), at 4th week and at 8th week of intervention
  Autoanalyzer Autoanalyzer Autoanalyzer
Lactic acid | At baseline and at 4th week of control condition; at baseline (before intervention), at 4th week and at 8th week of intervention
  Measured using photometry
Erythrocyte sedimentation rate (ESR) | At baseline and at 4th week of control condition; at baseline (before intervention), at 4th week and at 8th week of intervention
  Wintrobe Method
γ-Glutamyltransferase (GGT) | At baseline and at 4th week of control condition; at baseline (before intervention), at 4th week and at 8th week of intervention
  Measured with commercial kit
Aspartate Aminotransferase (AST) | At baseline and at 4th week of control condition; at baseline (before intervention), at 4th week and at 8th week of intervention
  Measured with commercial kit
Alanine Aminotransferase (ALT) | At baseline and at 4th week of control condition; at baseline (before intervention), at 4th week and at 8th week of intervention
  Measured with commercial kit
Sit and reach flexibility test for the hamstrings muscles and lower back | At baseline and at 4th week of control condition; at baseline (before intervention), at 4th week and at 8th week of intervention
  Each participant sits on the floor with legs stretched out straight ahead, reaches out and holds that position for at 1-2 seconds while the distance is recorded.
Grip strength | At baseline and at 4th week of control condition; at baseline (before intervention), at 4th week and at 8th week of intervention
  Handgrip strength test
Number of push-ups performed in one minute | At baseline and at 4th week of control condition; at baseline (before intervention), at 4th week and at 8th week of intervention
Number of sit-ups performed until exhaustion | At baseline and at 4th week of control condition; at baseline (before intervention), at 4th week and at 8th week of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yannis Theodorakis, PhD, Study Chair — University of Thessaly

IPD SHARING:
Plan to Share IPD: No